CLINICAL TRIAL: NCT04948567
Title: Efficacy of Split-dose of Oral Magnesium Sulfate Solution for Bowel Preparation in Elderly Patients
Brief Title: Efficacy of Split-dose of Oral MMS for Bowel Preparation in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, associated professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY20170119-2
Record Dates: First submitted 2021-05-27; First posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-05

CONDITIONS: Colonic Adenoma; Bowel Preparation
Keywords: bowel preparation; Oral magnesium sulfate solution; polyethylene glycol solution

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- split-dose of Magnesium Sulfate solution (Experimental): Those assigned to MSS group were instructed to take 30ml of 50% magnesium sulfate solution and then drink 600ml water on the evening before colonoscopy. 70ml of 50% MMS and then 1500ml water was taken at least 4 hours before procedure on the colonoscopy day.
  Interventions: Other: split-dose of Magnesium Sulfate solution
- split-dose of PEG (Placebo Comparator): Patients in PEG group were instructed to take first dose of 1.5L PEG on the evening before colonoscopy and take the second dose of 1.5L PEG at least 4 hours before the colonoscopy procedure on the morning.
  Interventions: Other: split-dose of PEG

INTERVENTIONS:
Other: split-dose of Magnesium Sulfate solution — purgative for bowel preparation
  Arms: split-dose of Magnesium Sulfate solution
Other: split-dose of PEG — purgative for bowel preparation
  Arms: split-dose of PEG

SUMMARY:
Adequate bowel preparation is critical for successful colonoscopy and a large volume of PEG was required for bowel preparation in patients undergoing colonoscopy. The investigators conducted a a prospective, randomized, controlled study to compare low dose of oral magnesium sulfate solution with high dose PEG. The investigators found that patients who took low dose of oral magnesium sulfate solution had similar bowel preparation quality to patients who took PEG,but accompanied with fewer adverse events and better tolerance.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent colonoscopy

Exclusion Criteria:

* known or suspected bowel stricture or obstruction;
* history of colorectal surgery;
* significant gastroparesis or gastric outlet obstruction;
* toxic colitis or megacolon;
* severe acute inflammatory bowel disease;
* active gastrointestinal bleeding;
* suspected or confirmed chronic renal insufficiency and heart illness;
* disturbance of electrolytes ;
* unable to provide informed consent

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1174 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
The rate of patients with adequate bowel preparation | 1 year
  Defined by each segmental BBPS≥2

SECONDARY OUTCOMES:
The rate of adenoma detection | 1 year
  The proportion of participants with at least one adenoma in each group
the numbers of patients with adverse events | 1 year
  eg. Vomiting, nausea, abdominal pain
The cecal intubation rate | 1 year
  The rate of colonoscopy reaching the cecum
The time of Cecal intubation | during procedure
  the time between the intubation and visualization of any of the following anatomic landmarks: ileocecal valve, appendiceal orifice, or terminal ileum
the time during Withdrawal phage | during procedure
  the inspection time from cecum to rectum

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Endoscopic center, Xijing Hospital of Digestive Diseases, Xi’an, Shanxi
  - Department of Gastroenterology, The Second Medical Center & National Clinical Research Center for Geriatric Diseases, Chinese PLA General Hospital,, Beijing

REFERENCES:
- [Derived] Ge F, Kang X, Wang Z, Zhu H, Liao L, Wang M, Jia J, Lou L, Guo X, Pan Y, Wan J. Low-dose of magnesium sulfate solution was not inferior to standard regime of polyethylene glycol for bowel preparation in elderly patients: a randomized, controlled study. Scand J Gastroenterol. 2023 Jan;58(1):94-100. doi: 10.1080/00365521.2022.2106154. Epub 2022 Aug 3. PMID 35920250